CLINICAL TRIAL: NCT00029770
Title: Chiropractic Care, Medication, and Self-Care for Neck Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Purpose: Treatment
Other Study IDs: R01AT000707-01 (NIH)
Record Dates: First submitted 2002-01-23; First posted 2002-01-24 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Manipulation, Chiropractic; Acetaminophen; Self Care; Anti-Inflammatory Agents, Non-Steroidal; acetaminophen, codeine drug combination

INTERVENTIONS:
Procedure: Chiropractic spinal manipulation
Drug: Acetaminophen
Behavioral: Self-care
Drug: Non-Steroidal anti-inflammatory drugs (NSAIDS)
Drug: Tylenol with codeine

SUMMARY:
This study will compare the effectiveness of chiropractic care, medications, and self-care on neck pain, a very common condition. The broad, long-term objective of this study is to identify effective therapies for neck pain sufferers and to increase understanding of neck pain conditions.

DETAILED DESCRIPTION:
Neck pain is very common, with considerable socioeconomic consequences. Although some therapies appear promising, there are too few randomized clinical trials of sufficient quality to support the use of one therapy over another. This is especially true for acute/subacute neck pain. Although commonly treated with prescription medications, neck pain sufferers are increasingly seeking relief through complementary and alternative medicine therapies, such as chiropractic spinal manipulation. Little is known, however about the short- and long-term relative efficacy of these therapies and how they compare to giving patients simple advice on self-care.

The broad, long-term objective of this research is to identify effective therapies for neck pain sufferers and to increase our understanding of neck pain conditions. This randomized, observer-blinded clinical trial is a unique collaborative effort by experienced chiropractic and medical researchers and will focus on patients with acute/subacute neck pain (<12 weeks duration). The study will determine the relative efficacy of chiropractic spinal manipulation, prescription medication, and self-care advice for neck pain in both the short term (after 6 weeks) and long term (after 52 weeks), using patient-rated neck pain as the main indicator of success.

ELIGIBILITY:
Exclusion Criteria:

* Pregnant women, due to use of diagnostic procedures (x-rays) and study treatments (NSAIDs and narcotic medications)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270
Dates: Start 2001-09; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Health Sciences University, Bloomington, Minnesota, United States

REFERENCES:
- [Derived] Bronfort G, Evans R, Anderson AV, Svendsen KH, Bracha Y, Grimm RH. Spinal manipulation, medication, or home exercise with advice for acute and subacute neck pain: a randomized trial. Ann Intern Med. 2012 Jan 3;156(1 Pt 1):1-10. doi: 10.7326/0003-4819-156-1-201201030-00002. PMID 22213489